CLINICAL TRIAL: NCT03297268
Title: Behavioral and Environmental Sensing and Intervention for Dementia Caregiver Empowerment
Brief Title: Behavioral and Environmental Sensing and Intervention
Acronym: BESI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: Carilion Clinic (Other); North Carolina Agriculture & Technical State University (Other)
Responsible Party: Sponsor
Other Study IDs: 0037457000; 1418622 (Other Grant/Funding Number: National Science Foundation)
Record Dates: First submitted 2017-09-20; First posted 2017-09-29 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Behavioral and Psychiatric Symptoms of Dementia; Dementia; Caregivers
Keywords: Dementia Caregiver Empowerment; Caregiver Burden; Agitation in Dementia; Environmental Sensors; Wearable Technology
MeSH Terms: conditions — Behavior; Dementia; Caregiver Burden; Aberrant Motor Behavior in Dementia | interventions — Methods

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Phase 1-Controlled Validation & Study Planning: Phase 1 is focused on refining and ultimately verifying BESI's basic sensing and notification functionality and validating BESI's environmental assessments in a controlled setting - namely the laboratory and homes of two healthy volunteers. This phase also serves to support further requirements gathering to refine BESI for community-based deployment. No interventions are delivered.
- Phase 2 - In-situ Validation and Ethnographic Analysis: Phase 2 starts the deployment of the technology within a community context, with the goals of validating the system's ability to assess agitation and environmental events in-situ and developing the cyber-sociophysical system models based on the dyad-specific relationship between agitation and the environment. A hybrid remote ethnographic methodology will be used, combining remote BESI measurement and caregiver diaries and a time-series design for the administration of the assessment battery.
- Phase 3 - Intervention with Home-Based Caregivers: Phase 3 is the intervention phase and the full realization of BESI. The goal is to employ the validated assessment capabilities and the developed modeling techniques to enable real-time, dyad-specific caregiver notifications that empower a caregiver to intervene with the PWD and/or environment before agitation escalation. In addition to validation of the BESI's ability to provide such appropriate notifications, Phase 3 will also serve as a pilot study about the effect that these notifications have on caregiver empowerment (as measured by self-efficacy) and the frequency and severity of PWD agitation, thus providing proof-of-concept for BESI's potential to improve dyad outcomes and motivating a larger-scale followup study to establish proof-of-practice.
  Interventions: Other: Intervention with Home-Based Caregivers

INTERVENTIONS:
Other: Intervention with Home-Based Caregivers — We will assess whether real-time notifications of potential agitation via a wearable wrist device improves caregiver self-efficacy.
  Other Names: Real-time caregiver notifications
  Groups: Phase 3 - Intervention with Home-Based Caregivers

SUMMARY:
This 3-phase research plan to employ Behavioral and Environmental Sensing and Intervention (BESI) will overcome the fundamental scientific barriers to realizing prediction of agitation episodes and detection early stages of dementia related agitation. The goal of which is empowering caregivers to intervene early and ultimately reduce agitation, thus reducing caregiver burden and extending aging-in-place and improving the associated quality-of-life and cost benefits.

DETAILED DESCRIPTION:
The dementia syndrome of Alzheimer's disease and other disorders is rapidly expanding due to the aging of society and the longevity of citizens. In its varying stages, care of the dementia syndrome requires differing sets of skills from the caregivers, and more skilled intervention is required as the disease progresses. These caregivers experience increased burden due to the challenges and stresses of caring. A recent systematic review of caregiver burden factors revealed dementia-related agitation to be the most prevalent factor leading caregivers to institutionalize community-dwelling loved ones with dementia. Tools that empower caregivers to proactively reduce the incidents and severity of agitation would reduce stress and increase self-efficacy, thereby extending aging-in-place and the associated quality-of-life and cost benefits.

This project proposes to develop, deploy, and evaluate such a tool and to address the fundamental scientific challenges to realizing the benefits of such a technology to caregivers and persons with dementia (PWD). The tool - BESI: Behavioral and Environmental Sensing and Intervention - will be an empowerment tool for caregivers of community-dwelling PWD. BESI comprises:

1. a system of body-worn inertial sensors and in-home acoustic, light, temperature, and motion sensors,
2. data analysis techniques to detect and assess agitation and environmental context from these sensor streams,
3. models for the relationship between agitation and the environment that are trained for each PWD-caregiver dyad based on a&b, and
4. automated real-time notifications to the caregiver based on b&c (e.g., detection of early agitation stages or of an environment (cumulative and/or instantaneous based on the models) that has led to agitation in the past), empowering the caregiver to intervene before agitation escalation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of dementia
* Living in one home for at least 2 months without hospitalization
* Caregiver seeking support for caregiving needs
* Have a stable caregiver
* Be able to provide consent or assent

Exclusion Criteria:

* Hospitalization in the last 2 months
* Multiple and inconsistent caregivers
* Living in multiple homes
* Unable to provide consent or assent
* No known dementia

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample of people with dementia living at home with unpaid caregivers.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Improved Caregiver Self-Efficacy | 30 days
  Increased scores on Revised Scale for Caregiver Self-Efficacy
Decreased Caregiver Burden | 30 days
  Zarit Burden Interview score lowered

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alzheimer's Association. 2016 Alzheimer's disease facts and figures. Alzheimers Dement. 2016 Apr;12(4):459-509. doi: 10.1016/j.jalz.2016.03.001. PMID 27570871
- [Background] Friedman EM, Shih RA, Langa KM, Hurd MD. US Prevalence And Predictors Of Informal Caregiving For Dementia. Health Aff (Millwood). 2015 Oct;34(10):1637-41. doi: 10.1377/hlthaff.2015.0510. PMID 26438738
- [Background] Cohen-Mansfield J, Billig N. Agitated behaviors in the elderly. I. A conceptual review. J Am Geriatr Soc. 1986 Oct;34(10):711-21. doi: 10.1111/j.1532-5415.1986.tb04302.x. PMID 3531296
- [Background] Cummings J, Mintzer J, Brodaty H, Sano M, Banerjee S, Devanand DP, Gauthier S, Howard R, Lanctot K, Lyketsos CG, Peskind E, Porsteinsson AP, Reich E, Sampaio C, Steffens D, Wortmann M, Zhong K; International Psychogeriatric Association. Agitation in cognitive disorders: International Psychogeriatric Association provisional consensus clinical and research definition. Int Psychogeriatr. 2015 Jan;27(1):7-17. doi: 10.1017/S1041610214001963. Epub 2014 Oct 14. PMID 25311499
- [Background] Cohen-Mansfield J, Marx MS, Rosenthal AS. A description of agitation in a nursing home. J Gerontol. 1989 May;44(3):M77-84. doi: 10.1093/geronj/44.3.m77. PMID 2715584
- [Background] Colombo M, Vitali S, Cairati M, Vaccaro R, Andreoni G, Guaita A. Behavioral and psychotic symptoms of dementia (BPSD) improvements in a special care unit: a factor analysis. Arch Gerontol Geriatr. 2007;44 Suppl 1:113-20. doi: 10.1016/j.archger.2007.01.017. PMID 17317443
- [Background] Steinberg M, Shao H, Zandi P, Lyketsos CG, Welsh-Bohmer KA, Norton MC, Breitner JC, Steffens DC, Tschanz JT; Cache County Investigators. Point and 5-year period prevalence of neuropsychiatric symptoms in dementia: the Cache County Study. Int J Geriatr Psychiatry. 2008 Feb;23(2):170-7. doi: 10.1002/gps.1858. PMID 17607801
- [Background] Sansoni J, Anderson KH, Varona LM, Varela G. Caregivers of Alzheimer's patients and factors influencing institutionalization of loved ones: some considerations on existing literature. Ann Ig. 2013 May-Jun;25(3):235-46. doi: 10.7416/ai.2013.1926. PMID 23598807
- [Background] Fonareva I, Oken BS. Physiological and functional consequences of caregiving for relatives with dementia. Int Psychogeriatr. 2014 May;26(5):725-47. doi: 10.1017/S1041610214000039. Epub 2014 Feb 10. PMID 24507463
- [Background] Mausbach BT, Chattillion EA, Roepke SK, Patterson TL, Grant I. A comparison of psychosocial outcomes in elderly Alzheimer caregivers and noncaregivers. Am J Geriatr Psychiatry. 2013 Jan;21(1):5-13. doi: 10.1016/j.jagp.2012.10.001. Epub 2013 Jan 2. PMID 23290198
- [Background] Epstein-Lubow G, Gaudiano B, Darling E, Hinckley M, Tremont G, Kohn R, Marino LJ Jr, Salloway S, Grinnell R, Miller IW. Differences in depression severity in family caregivers of hospitalized individuals with dementia and family caregivers of outpatients with dementia. Am J Geriatr Psychiatry. 2012 Sep;20(9):815-9. doi: 10.1097/JGP.0b013e318235b62f. PMID 21997604
- [Background] Bankole A, Anderson M, Smith-Jackson T, Knight A, Oh K, Brantley J, Barth A, Lach J. Validation of noninvasive body sensor network technology in the detection of agitation in dementia. Am J Alzheimers Dis Other Demen. 2012 Aug;27(5):346-54. doi: 10.1177/1533317512452036. PMID 22815084
- [Background] Rowe M, Lane S, Phipps C. CareWatch: A Home Monitoring System for Use in Homes of Persons With Cognitive Impairment. Top Geriatr Rehabil. 2007 Jan 1;23(1):3-8. doi: 10.1097/00013614-200701000-00003. PMID 20454554
- [Background] Sacco G, Joumier V, Darmon N, Dechamps A, Derreumaux A, Lee JH, Piano J, Bordone N, Konig A, Teboul B, David R, Guerin O, Bremond F, Robert P. Detection of activities of daily living impairment in Alzheimer's disease and mild cognitive impairment using information and communication technology. Clin Interv Aging. 2012;7:539-49. doi: 10.2147/CIA.S36297. Epub 2012 Dec 4. PMID 23271900
- [Background] Perlman CM, Hirdes JP. The aggressive behavior scale: a new scale to measure aggression based on the minimum data set. J Am Geriatr Soc. 2008 Dec;56(12):2298-303. doi: 10.1111/j.1532-5415.2008.02048.x. PMID 19093929
- [Background] Hall GR, Gerdner LA, Zwygart-Stauffacher M, et al: Principles of nonpharmacological management: Caring for people with Alzheimer's disease using a conceptual model. Psychiatric Annals 1995; 25(7):432-440
- [Background] Smith M, Gerdner LA, Hall GR, Buckwalter KC. History, development, and future of the progressively lowered stress threshold: a conceptual model for dementia care. J Am Geriatr Soc. 2004 Oct;52(10):1755-60. doi: 10.1111/j.1532-5415.2004.52473.x. PMID 15450057
- [Background] Gerdner LA, Buckwalter KC, Hall GR: Temporal patterning of agitation and stressors associated with agitation: Case profiles to illustrate the Progressively Lowered Stress Threshold model. Journal of the American Psychiatric Nurses Association 2005; 11(4):215-222
- [Background] Kaufer DI, Cummings JL, Ketchel P, Smith V, MacMillan A, Shelley T, Lopez OL, DeKosky ST. Validation of the NPI-Q, a brief clinical form of the Neuropsychiatric Inventory. J Neuropsychiatry Clin Neurosci. 2000 Spring;12(2):233-9. doi: 10.1176/jnp.12.2.233. PMID 11001602
- [Background] Sclan SG, Reisberg B. Functional assessment staging (FAST) in Alzheimer's disease: reliability, validity, and ordinality. Int Psychogeriatr. 1992;4 Suppl 1:55-69. doi: 10.1017/s1041610292001157. PMID 1504288
- [Background] Teng EL, Chui HC. The Modified Mini-Mental State (3MS) examination. J Clin Psychiatry. 1987 Aug;48(8):314-8. PMID 3611032
- [Background] Morris JC. The Clinical Dementia Rating (CDR): current version and scoring rules. Neurology. 1993 Nov;43(11):2412-4. doi: 10.1212/wnl.43.11.2412-a. No abstract available. PMID 8232972
- [Background] Alexopoulos GS, Abrams RC, Young RC, Shamoian CA. Cornell Scale for Depression in Dementia. Biol Psychiatry. 1988 Feb 1;23(3):271-84. doi: 10.1016/0006-3223(88)90038-8. PMID 3337862
- [Background] Orme JG, Reis J, Herz EJ. Factorial and discriminant validity of the Center for Epidemiological Studies Depression (CES-D) scale. J Clin Psychol. 1986 Jan;42(1):28-33. doi: 10.1002/1097-4679(198601)42:13.0.co;2-t. PMID 3950011
- [Background] Steffen AM, McKibbin C, Zeiss AM, Gallagher-Thompson D, Bandura A. The revised scale for caregiving self-efficacy: reliability and validity studies. J Gerontol B Psychol Sci Soc Sci. 2002 Jan;57(1):P74-86. doi: 10.1093/geronb/57.1.p74. PMID 11773226
- [Background] Bedard M, Molloy DW, Squire L, Dubois S, Lever JA, O'Donnell M. The Zarit Burden Interview: a new short version and screening version. Gerontologist. 2001 Oct;41(5):652-7. doi: 10.1093/geront/41.5.652. PMID 11574710
- [Background] MAHONEY FI, BARTHEL DW. FUNCTIONAL EVALUATION: THE BARTHEL INDEX. Md State Med J. 1965 Feb;14:61-5. No abstract available. PMID 14258950
- [Background] Duffy L, Gajree S, Langhorne P, Stott DJ, Quinn TJ. Reliability (inter-rater agreement) of the Barthel Index for assessment of stroke survivors: systematic review and meta-analysis. Stroke. 2013 Feb;44(2):462-8. doi: 10.1161/STROKEAHA.112.678615. Epub 2013 Jan 8. PMID 23299497
- [Background] Logsdon RG, Gibbons LE, McCurry, et al: Quality of life in Alzheimer's disease: Patient and caregiver reports. Journal of Mental Health and Ageing 1999; 5:21-32
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Grissom RJ. Heterogeneity of variance in clinical data. J Consult Clin Psychol. 2000 Feb;68(1):155-65. doi: 10.1037//0022-006x.68.1.155. PMID 10710850
- [Background] Jeste DV, Palmer BW, Appelbaum PS, Golshan S, Glorioso D, Dunn LB, Kim K, Meeks T, Kraemer HC. A new brief instrument for assessing decisional capacity for clinical research. Arch Gen Psychiatry. 2007 Aug;64(8):966-74. doi: 10.1001/archpsyc.64.8.966. PMID 17679641
- [Background] Hurd MD, Martorell P, Delavande A, Mullen KJ, Langa KM. Monetary costs of dementia in the United States. N Engl J Med. 2013 Apr 4;368(14):1326-34. doi: 10.1056/NEJMsa1204629. PMID 23550670
- See also: Wearable device used in BESI — http://www.pebble.com